CLINICAL TRIAL: NCT01118325
Title: A Randomised, Double-Blind, Parallel Group, Asian, Multicenter Study, to Assess Pharmacokinetic and Pharmacodynamic Profile of 2 Doses of Ticagrelor on Top of Low Dose Acetyl Salicylic Acid (ASA) Therapy on Platelet Aggregation in Japanese and Asian Patients With Stable Coronary Artery Disease
Brief Title: An Asian Study to Assess the Properties and Profile of Ticagrelor in Patients With Stable Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5130C00065
Record Dates: First submitted 2010-04-30; First posted 2010-05-06 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Stable Coronary Artery Disease
Keywords: Stable Coronary Artery Disease; Platelet Aggregation
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AZD6140 45 mg bd (Experimental)
  Interventions: Drug: ticagrelor
- AZD6140 90 mg bd (Experimental)
  Interventions: Drug: ticagrelor
- Clopidogrel 75 mg od (Active Comparator)
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: ticagrelor — Drug oral treatment
  Arms: AZD6140 45 mg bd; AZD6140 90 mg bd
Drug: clopidogrel — Drug oral treatment
  Arms: Clopidogrel 75 mg od

SUMMARY:
The purpose of the study is to determine the drug characteristics of Ticagrelor, and to determine if 4 weeks treatment will reduce the blood clotting.

ELIGIBILITY:
Inclusion Criteria:

* Any Percutaneous Coronary Intervention, more than 3 months prior to randomization
* Previous documented acute coronary syndrome (ACS), more than 3 months prior to randomisation
* Treatment with ASA

Exclusion Criteria:

* ACS, transient ischemic attack (TIA), or Stroke within the 3 months prior to randomisation
* Known concurrent disease of stroke or TIA with atrial fibrillation
* Persons who are being treated with blood clotting agents that cannot be stopped

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C. Fox, MD, Study Director — AstraZeneca
Locations (13):
- Japan (11):
  - Research Site, Miyaodai, Fukuoka
  - Research Site, Sapporo, Hokkaido
  - Research Site, Toride-shi, Ibaraki
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Naha, Okinawa
  - Research Site, Osaka, Osaka
  - Research Site, Kusatsu-shi, Shiga
  - Research Site, Komatsushima-shi, Tokushima
  - Research Site, Shinagawa-ku, Tokyo
- Philippines (2):
  - Research Site, Davao City
  - Research Site, Quezon City

REFERENCES:
- [Background] Hiasa Y, Teng R, Emanuelsson H. Pharmacodynamics, pharmacokinetics and safety of ticagrelor in Asian patients with stable coronary artery disease. Cardiovasc Interv Ther. 2014 Oct;29(4):324-33. doi: 10.1007/s12928-014-0277-1. Epub 2014 Jun 17. PMID 24935072
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=374&filename=CSR-D5130C00065.pdf
- See also: CSR-D5130C00065.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=374&filename=CSR-D5130C00065.pdf
- See also: D5130C00065_CSP_redacted_17_Oct_2013 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=374&filename=D5130C00065_CSP_Redacted_17_Oct_2013.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 146 patients were enrolled at 15 sites from 2 countries (Japan and Philippines). The study period was from April 2010 to March 2011. In total, 139 subjects were randomised and received the investigational product. Most subjects completed the study but 2 Japanese patients discontinued due to an AE during the 4 weeks treatment period.
Groups:
- AZD6140 45 mg bd: AZD6140 45 mg twice daily
- AZD6140 90 mg bd: AZD6140 90 mg twice daily
- Clopidogrel 75 mg od: Clopidogrel 75 mg once daily
Period: Overall Study
Arm/Group | AZD6140 45 mg bd | AZD6140 90 mg bd | Clopidogrel 75 mg od
Started | 50 | 43 | 46
Completed | 49 | 43 | 45
Not Completed | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD6140 45 mg bd | AZD6140 90 mg bd | Clopidogrel 75 mg od | Total
Number analyzed (Participants) | 50 | 43 | 46 | 139
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (11) | 64 (9) | 64 (10) | 63 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 8 | 15
  Male | 46 | 40 | 38 | 124
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 42 | 35 | 40 | 117
  Non-Japanese | 8 | 8 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Inhibition of Platelet Aggregation(IPA) Final Extent at 2 Hours Post Dose on Week 4 in Japanese Patients
Description: Final extent IPA from pre-dose baseline was calculated using the following formula for Adenosine Diphosphate (ADP)-induced platelet aggregation:
  Percentage Inhibition = 100% x (PAs - PA) / (PAs) Platelet Aggregation (PA) was the mean response at the given post dose time point and PAs was the mean response at pre dose baseline. Percentage inhibition was restricted to the closed interval [0,100]; any data falling outside this range was truncated to the appropriate limit.
Time Frame: Week 4
Population: Only Japanese participants who had IPA data at Week 4 were considered in this analysis. Arm AZD6140 90 mg bd includes one non-Japanese participant resident in Japan
Measure: Mean (Standard Deviation); unit: percentage inhibition
Groups:
- AZD6140 45 mg bd: AZD6140 45 mg twice daily in Japanese patients
- AZD6140 90 mg bd: AZD6140 90 mg twice daily in Japanese patients
Arm/Group | AZD6140 45 mg bd | AZD6140 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 41 | 36 | 39
percentage inhibition | 64.5 (14.8) | 73.0 (14.2) | 38.9 (20.7)

2. Primary Outcome: IPA Final Extent at 4 Hours Post Dose on Week 4 in Japanese Patients
Description: Final extent IPA from pre-dose baseline was calculated using the following formula for ADP-induced platelet aggregation:
  Percentage Inhibition = 100% x (PAs - PA) / (PAs) PA was the mean response at the given post dose time point and PAs was the mean response at pre dose baseline. Percentage inhibition was restricted to the closed interval [0,100]; any data falling outside this range was truncated to the appropriate limit.
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage inhibition
Arm/Group | AZD6140 45 mg bd | AZD6140 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 41 | 36 | 39
percentage inhibition | 67.3 (15.6) | 73.2 (15.1) | 43.7 (20.6)

3. Primary Outcome: IPA Final Extent at 8 Hours Post Dose on Week 4 in Japanese Patients
Description: as for outcome 2
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage inhibition
Arm/Group | AZD6140 45 mg bd | AZD6140 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 41 | 36 | 39
percentage inhibition | 62.7 (17.7) | 68.6 (16.0) | 42.5 (20.2)

4. Primary Outcome: IPA Final Extent at 12 Hours Post Dose on Week 4 in Japanese Patients
Description: as for outcome 2
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage inhibition
Groups:
- Arm 1 - AZD6140 45 mg bd: AZD6140 45 mg twice daily
Arm/Group | Arm 1 - AZD6140 45 mg bd | AZD6140 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 41 | 36 | 39
percentage inhibition | 56.9 (20.9) | 66.8 (20.1) | 41.8 (21.7)

5. Primary Outcome: IPA Final Extent at 24 Hours Post Dose on Week 4 in Japanese Patients
Description: as for outcome 2
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage inhibition
Arm/Group | AZD6140 45 mg bd | AZD6140 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 41 | 36 | 39
percentage inhibition | 46.2 (23.3) | 59.1 (20.3) | 38.0 (20.5)

6. Secondary Outcome: AZD6140 (Cmax) at Week 4
Description: Maximum plasma AZD6140 concentration
Time Frame: Week 4
Population: Only Japanese participants who had IPA data at Week 4 were considered in this analysis
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- AZD6140 45 mg bd in Japanese Patients: AZD6140 45 mg twice daily in Japanese patients
- AZD6140 45 mg bd in Non-Japanese Patients: AZD6140 45 mg twice daily in non-Japanese patients
- AZD6140 90 mg bd in Japanese Patients: AZD6140 90 mg twice daily in Japanese patients
- AZD6140 90 mg bd in Non-Japanese Patients: AZD6140 90 mg twice daily in non-Japanese patients
Arm/Group | AZD6140 45 mg bd in Japanese Patients | AZD6140 45 mg bd in Non-Japanese Patients | AZD6140 90 mg bd in Japanese Patients | AZD6140 90 mg bd in Non-Japanese Patients
Number analyzed (Participants) | 38 | 8 | 33 | 7
ng/mL | 422 (230) | 341 (370) | 931 (442) | 1380 (343)

7. Secondary Outcome: AZD6140 (AUC0-tau) at Week 4
Description: Area under the plasma concentration curve of AZD6140 from time zero to dosing interval
Time Frame: Week 4
Population: In total 7 Japanese patients (4 patients in 45 mg and 3 patients in 90 mg) were excluded from the PK analysis set since PK samples of these patients were discarded due to a database set-up issue at the central laboratory.
Measure: Geometric Mean (Standard Deviation); unit: ng.h/mL
Groups:
- AZD6140 45 mg bd in Non-Japanese Patients: AZD6140 90 mg twice daily in non-Japanese patients
- AZD6140 90 mg bd in Non-Japanese Patients: AZD6140 45 mg twice daily in non-Japanese patients
Arm/Group | AZD6140 45 mg bd in Japanese Patients | AZD6140 45 mg bd in Non-Japanese Patients | AZD6140 90 mg bd in Japanese Patients | AZD6140 90 mg bd in Non-Japanese Patients
Number analyzed (Participants) | 38 | 8 | 33 | 7
ng.h/mL | 3050 (1940) | 2930 (3740) | 6080 (2600) | 10900 (2790)

8. Secondary Outcome: AZD6140 (Tmax) at Week 4
Description: Time to reach peak or maximum concentration of AZD6140 following AZD6140 administration
Time Frame: Week 4
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | AZD6140 45 mg bd in Japanese Patients | AZD6140 45 mg bd in Non-Japanese Patients | AZD6140 90 mg bd in Japanese Patients | AZD6140 90 mg bd in Non-Japanese Patients
Number analyzed (Participants) | 38 | 8 | 33 | 7
hour | 2.0 [1.9 to 4.0] | 4.0 [2.0 to 4.0] | 2.0 [1.9 to 4.1] | 4.0 [2.0 to 4.1]

9. Secondary Outcome: AR-C124910XX (Cmax) at Week 4
Description: Maximum plasma concentration of AZD6140 drug metabolite AR-C124910XX
Time Frame: Week 4
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- AZD6140 45mg bd in Non-Jpanese Patients: AZD6140 45 mg twice daily in non-Japanese patients
- AZD6140 90 mg bd in Non-Jpanese Patients: AZD6140 90 mg twice daily in non-Japanese patients
Arm/Group | AZD6140 45 mg bd in Japanese Patients | AZD6140 45mg bd in Non-Jpanese Patients | AZD6140 90 mg bd in Japanese Patients | AZD6140 90 mg bd in Non-Jpanese Patients
Number analyzed (Participants) | 38 | 8 | 33 | 7
ng/mL | 135 (53.3) | 101 (72.4) | 326 (139) | 381 (192)

10. Secondary Outcome: AR-C124910XX (AUC0-tau) at Week 4
Description: Area under the plasma concentration curve of AZD6140 drug metabolite AR-C124910XX from time zero to dosing interval
Time Frame: Week 4
Population: as for outcome 7
Measure: Geometric Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | AZD6140 45 mg bd in Japanese Patients | AZD6140 45 mg bd in Non-Japanese Patients | AZD6140 90 mg bd in Japanese Patients | AZD6140 90 mg bd in Non-Japanese Patients
Number analyzed (Participants) | 38 | 8 | 33 | 7
ng.h/mL | 1180 (490) | 954 (741) | 2720 (915) | 3380 (1580)

11. Secondary Outcome: AR-C124910XX (Tmax) at Week 4
Description: Time to reach peak or maximum concentration of AZD6140 drug metabolite AR-C124910XX following AZD6140 administration
Time Frame: Week 4
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | AZD6140 45 mg bd in Japanese Patients | AZD6140 45 mg bd in Non-Japanese Patients | AZD6140 90 mg bd in Japanese Patients | AZD6140 90 mg bd in Non-Japanese Patients
Number analyzed (Participants) | 38 | 8 | 33 | 7
hour | 4.0 [1.9 to 11.9] | 4.0 [2.0 to 8.0] | 2.1 [1.9 to 8.0] | 2.0 [2.0 to 4.0]

ADVERSE EVENTS:
Arm/Group | AZD6140 45 mg bd | AZD6140 90 mg bd | Clopidogrel 75 mg od
Serious Adverse Events (participants affected / at risk) | 2/50 | 1/43 | 0/46
Other Adverse Events (participants affected / at risk) | 13/50 | 23/43 | 9/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD6140 45 mg bd (N=50) | AZD6140 90 mg bd (N=43) | Clopidogrel 75 mg od (N=46)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
LIP AND/OR ORAL CAVITYCANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD6140 45 mg bd (N=50) | AZD6140 90 mg bd (N=43) | Clopidogrel 75 mg od (N=46)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 9 | 9 | 3
Nasopharyngitis (Infections and infestations) | 1 | 7 | 3
Abdominal discomfort (Gastrointestinal disorders) | 2 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less